CLINICAL TRIAL: NCT03809728
Title: IDENTIFICATION OF PROGNOSTIC AND PREDICTIVE BIOMARKERS OF NATURAL HISTORY AND RESPONSE TO BIOTHERAPIES IN INFLAMMATORY BOWEL DISEASE : i-BANK
Brief Title: IDENTIFICATION OF PROGNOSTIC AND PREDICTIVE BIOMARKERS IN INFLAMMATORY BOWEL DISEASE
Acronym: i-BANK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Laurent PEYRIN-BIROULET, Doctor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSS 2018 / I-BANK-GERMAIN / MS
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBD patients (Other): All patients with an established Crohn's disease or ulcerative colitis
  Interventions: Procedure: endoscopic biopsy; Procedure: samples of the oral cavity; Procedure: Samples of the resected specimen

INTERVENTIONS:
Procedure: endoscopic biopsy — Per-endoscopic biopsies
Procedure: samples of the oral cavity — 7 samples of the oral cavity with a swab
Procedure: Samples of the resected specimen — if patient has to undergo a digestive resection as part of his standard management, samples of the pathological area and samples at the end of the resection will be realised

SUMMARY:
Interventional study of a group of patients with an inflammatory bowel disease (IBD; Crohn's disease (CD) or ulcerative colitis (UC)) to identify predictive and prognostic biomarkers of natural history and response to biotherapies.

DETAILED DESCRIPTION:
Percentage of primary responders who haven't lost response to biotherapies during follow-up (anti-TNF, ustekinumab, vedolizumab).

Response to treatment will be evaluated using objective criteria for measuring intestinal inflammation: endoscopic remission (endoscopic biopsy and surgical specimens), radiological (MRI), and / or biological (CRP, fecal calprotectin) .

Response to therapy rates will be correlated with genomic, epigenomic, and microbiota data stratified by major environmental factors (nutrition, tobacco, physical activity).

ELIGIBILITY:
Inclusion Criteria:

* Age>=18 years
* Patients with an established diagnosis of CD or UC (clinical, biological, radiological, endoscopic or histologic criteria)
* Patients >=45 kg
* Affiliated member of the Social Security system

Exclusion Criteria:

* Patients with an undetermined colitis
* Patients with a non established diagnosis of CD
* Women of childbearing age without a method of contraception
* Persons covered by articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code
* Pregnant women, breastfeeding women

  -- Age < 18 years
* Persons under legal protection
* Person who does not have the capacity to consent
* Persons under the age of 18 years who are deprived of their liberty by decision of a judicial or administrative authority (articles L. 3212-1 and L. 3213-1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2034-12-10 (Estimated); Study Completion 2034-12-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have lost response to biotherapies (anti-TNF, ustekinumab, vedolizumab). | 5 years

SECONDARY OUTCOMES:
Proportion of patients who underwent surgery | 5 years
Post-operative morbidity rates in IBD | 5 years
Surgical recurrent rate in Crohn's disease | 5 years
Proportion of patients with a destruction of the intestinal wall in CD (abscess, fistula) | 5 years
Proportion of patients developing a cancer | 5 years
Readmission rates for acute severe colitis or ileitis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Adeline GERMAIN, MD, PhD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided